CLINICAL TRIAL: NCT05515783
Title: 68Ga-FAP-RGD PET/CT : Dosimetry and Preliminary Clinical Translational Studies in Cancer Patients
Brief Title: 68Ga-FAP-RGD PET/CT : Dosimetry and Preliminary Clinical Translational Studies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-FAP-RGD
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part I: safety, tolerability, biodistribution and dosimetry (Experimental): PET imaging will begin at 30s (30s/bed), 15min (1min/bed), 30min (2 min/bed), 60min (2 min/bed) and 120min (2 min/bed) after injection
  Interventions: Drug: 68Ga-FAP-RGD
- Part II: diagnostic efficacy (Experimental): Participants with various types of cancer will have PET imaging 50-100 minutes after injection of 68Ga-FAP-RGD and another agent (68Ga-FAPI-02 or 18F-FDG).
  Interventions: Drug: 68Ga-FAP-RGD

INTERVENTIONS:
Drug: 68Ga-FAP-RGD — The dose will be 4-7mCi given intravenously.
  Arms: Part I: safety, tolerability, biodistribution and dosimetry
Drug: 68Ga-FAP-RGD — 68Ga-FAP-CHX, the dose will be 0.05 (mCi / kg) given intravenously at a single time prior to imaging. 68Ga-FAPI-02, the dose will be 1.8 (MBq /kg) given intravenously at a single time prior to imaging; 18F-FDG, the dose will be 3.7 (MBq / kg) given intravenously at a single time prior to imaging.
  Arms: Part II: diagnostic efficacy

SUMMARY:
As an new dual targeting PET radiotracer, 68Ga-FAP-RGD is promising as an excellent imaging agent applicable to various cancers. In this study, we observed the safety, biodistribution and radiation dosimetry of 68Ga-FAP-RGD in patients with various types of cancer and compared them with the results of 68Ga-FAPI-02 or 18F-FDG imaging to evaluate the dosimetric characteristics and diagnostic efficacy of 68Ga-FAP-RGD.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is highly expressed in the stroma of a variety of human cancers and is therefore considered promising for guiding targeted therapy. The recent development of quinoline-based PET tracers that act as FAP inhibitors (FAPIs) demonstrated promising results preclinically and already in a few clinical cases. Integrin αvβ3 is restrictedly expressed on angiogenic blood vessels and tumour cells. It plays a key role in angiogenesis for tumour growth and metastasis. RGD peptide can specifically recognise the integrin αvβ3, which serves as targeted molecular for anti-angiogenesis strategies. 68Ga-FAP-RGD is a novel dual targeting tracers. The present study aimed to evaluate the biodistribution, pharmacokinetics, and dosimetry of 68Ga-FAP-RGD, and performed a head-to-head comparison with 68Ga-FAPI-02 or 18F-FDG PET/CT scans in patients with various cancers.

ELIGIBILITY:
Inclusion Criteria:

* Various solid tumors with available histopathological findings
* Signed informed consent

Exclusion Criteria:

* pregnant or lactational women
* who suffered from severe hepatic and renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Human biodistribution | From right after tracer injection to 2-hours post-injection
  reported as relative uptake values per organ at 30s, 15min, 30min, 60min and 120 min per individual subject and as a mean over all subjects (Part I)
Human dosimetry | From right after tracer injection to 2-hours post-injection
  radiation dose to individual organs and the equivalent dose for the whole body of each subject and as a mean over all subjects (Part I). Dosimetry will be calculated using the Hybrid-Dosimetry software.
Standard uptake value (SUV) | Up to 2 weeks
  Determination of SUV for detected lesions and discernible organs of 68Ga-FAP-RGD and 68Ga-FAPI-02 or 18F-FDG
Lesion numbers | Up to 2 weeks
  Determination of lesion numbers of 68Ga-FAP-RGD and 68Ga-FAPI-02 or 18F-FDG
the sensitivity of 68Ga-FAP-RGD PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the sensitivity of 68Ga-FAP-RGD PET/CT was evaluated.
the specificity of 68Ga-FAP-RGD PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the specificity of 68Ga-FAP-RGD PET/CT was evaluated.
the accuracy of 68Ga-FAP-RGD PET/CT | Up to 2 weeks
  compared with pathology or composite imaging, the accuracy of 68Ga-FAP-RGD PET/CT was evaluated.

SECONDARY OUTCOMES:
Count of participants with treatment emergent adverse events | Up to 3 days
  The frequency and severity of treatment emergent adverse events following 68Ga-FAP-RGD injection will be descriptively reported as classified and graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Study Chair — The First Affiliated Hospital, Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Zheng S, Zang J, Shao Z, Tu D, Liu Q, Chen X, Miao W, Zhang J. [68Ga]Ga-LNC1007 versus 2-[18F]FDG in the evaluation of patients with metastatic differentiated thyroid cancer: a head-to-head comparative study. Eur J Nucl Med Mol Imaging. 2025 Jan;52(2):683-692. doi: 10.1007/s00259-024-06930-4. Epub 2024 Oct 15. PMID 39404790
- [Derived] Zang J, Lin R, Wen X, Wang C, Zhao T, Jakobsson V, Yang Y, Wu X, Guo Z, Chen X, Zhang J, Miao W. A Head-to-Head Comparison of 68Ga-LNC1007 and 2-18F-FDG/68Ga-FAPI-02 PET/CT in Patients With Various Cancers. Clin Nucl Med. 2023 Oct 1;48(10):861-868. doi: 10.1097/RLU.0000000000004820. Epub 2023 Sep 2. PMID 37682601